CLINICAL TRIAL: NCT05547711
Title: Prediction and Validation of Unipolar Depression With Psychosocial-somatic Markers in a Naturalistic Cohort Recruited in an Outpatient Setting
Acronym: POKAL-PSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julia Eder (Other)
Responsible Party: Sponsor-Investigator, Julia Eder, Associate Physician, LMU Klinikum
Organization: LMU Klinikum (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22-0637; DFG-GRK 2621 POKAL (Other Grant/Funding Number: Prof. Dr.med. Jochen Gensichen); DRKS00030203 (Other: German Clinical Trials Register)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Depressive Disorder; Depression; Depressive Symptoms; Depressive Episode; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: At inclusion mentally healthy and patients with a depression are monitored for five years. After study inclusion participants will be seen after four weeks and then annually for five years.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with depression (Active Comparator)
  Interventions: Diagnostic Test: drawing blood
- Healthy controls (Active Comparator)
  Interventions: Diagnostic Test: drawing blood

INTERVENTIONS:
Diagnostic Test: drawing blood — drawing blood annually measurement of heartrate variability annually determine weight with a bioimpedance scale
  Other Names: bioimpedance scale; measurement of heartrate variability

SUMMARY:
The POKAL-PSY project is a study that monitors participants for five years. The goal of the study is to identify distinguishable subtypes of depression on the basis of biomarkers and to gain insight into their prognostic significance.

ELIGIBILITY:
Inclusion Criteria:

* (PHQ>8) if depressed
* Subjects of any sex aged between 18-70
* Sufficient ability to speak and understand the german language
* Ability to understand and sign the informed consent form

Exclusion Criteria:

* Cognitive impairment that interferes with reliable completion of questionnaires or answering questions
* Presence of manic episode, bipolar disorder, Schizophrenia or schizoaffective disorder (as well as other diseases in the F2 domain in the ICD), active eating disorder, active drug or alcohol dependence syndrome
* Presence of uncontrolled systemic disease (e.g. autoimmune disease), uncontrolles somatic (other than metabolic or cardiovascular)/ neurologic diseases, current or recent (last month) physical trauma
* Patient with acute suicidal ideation
* known deficiency of alpha-1-antitrypsin
* pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2032-10-15 (Estimated)

PRIMARY OUTCOMES:
Changes in GAF | 4 Weeks
Changes in MADRS | 4 Weeks
Alpha-1-Antitrypsin | 1 year
IGF-1 | 1 year
weight | 1 year

SECONDARY OUTCOMES:
Changes in GAF | 5 years
Changes in MADRS | 5 years
alpha-1-Antitrypsin | 5 years
IGF-1 | 5 years
weight | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital LMU, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be completely anonymised before conducting statistical analysis. First data will be shared within the graduate college.
  After fist publications other researches can use the data upon reasonable request
Supporting Information: Study Protocol
Time Frame: will be determined
Access Criteria: proposal

REFERENCES:
- See also: POKAL Website — https://pokal-kolleg.de/